CLINICAL TRIAL: NCT04304248
Title: A Phase II Study of Neoadjuvant Toripalimab Plus Platinum-based Doublet for Potentially Resectable Stage III Non-small Cell Lung Cancer
Brief Title: Neoadjuvant Toripalimab Plus Platinum-based Doublet for Stage III Non-small Cell Lung Cancer
Acronym: NeoTAP01
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hao Long (Other)
Responsible Party: Sponsor-Investigator, Hao Long, Prof., Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC B2019-116-01
Record Dates: First submitted 2020-03-09; First posted 2020-03-11 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non small cell lung cancer; neoadjuvant; chemo-immunotherapy; Toripalimab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Albumin-Bound Paclitaxel; Carboplatin; toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant chemo-immunotherapy (Experimental): Neoadjuvant treatment (Albumin-bound paclitaxel + carboplatin + toripalimab) will start within 1-3 days from enrollment at 21-day (+/-3 days) intervals (Q3W) prior to surgery. Before surgery a tumor assessment will be done to exclude evidence of progression. Patients with radiographically stable disease or partial response may be considered for operation.
  Surgery: Surgery must be done within the 3rd to 4th week (+7 days) from day 21 cycle 3 of neoadjuvant treatment.
  Interventions: Drug: Albumin-bound paclitaxel, Carboplatin, Toripalimab

INTERVENTIONS:
Drug: Albumin-bound paclitaxel, Carboplatin, Toripalimab — Eligible patients will receive Toripalimab 240mg + Albumin-bound paclitaxel 260mg/m2 + Carboplatin AUC5 for 3 cycles every 21 days (+/-3 days) as neoadjuvant treatment

SUMMARY:
This is an open-label, single-arm, phase II, multi-center clinical trial. Thirty patients will be enrolled in this trial to investigate the pathological complete response rate defined as the absence of residual tumor in lung and lymph nodes treated by chemo-immunotherapy.

DETAILED DESCRIPTION:
This is an open-label, single-arm, phase II, multi-center clinical trial. Eligible patients will receive Toripalimab 240mg + Albumin-bound paclitaxel 260mg/m2 + Carboplatin AUC5 for 3 cycles every 21 days (+/-3 days) as neoadjuvant treatment followed by surgery 3-4 weeks after the last dose of chemo-immunotherapy.

The primary objective is major pathologic response (MPR), defined as less than 10% tumor cells in the pathologically resected specimen. Patient accrual is expected to be completed within 18 months excluding a run-in-phase of 3 months. Patients will be followed 3 years after surgery. The study will end once survival follow-up has concluded.

ELIGIBILITY:
Inclusion Criteria:

1. Previously untreated patients with histologically- or cytologically- documented NSCLC who present stage IIIA disease (according to 8th version of the International Association for the Study of Lung Cancer Staging Manual in Thoracic Oncology) and also, potentially resectable locally advanced NSCLC patients' stage IIIB with T3N2 disease according to 8th edition can be included.

   PET/CT including IV contrast (CT of diagnostic quality) will be performed at baseline (28 days +10 before randomization);
2. Tumor should be EGFR wild-type or EML4-ALK negative;
3. Tumor should be considered resectable before study entry by a multidisciplinary team;
4. ECOG (Performance status) 0-1;
5. Screening laboratory values must meet the following criteria and should be obtained within 14 days prior to randomization.

   i. Neutrophils ≥ 1500×109/L ii. Platelets ≥ 100 x×109/L iii. Hemoglobin > 9.0 g/dL iv. Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 40 mL/min v. AST/ALT ≤ 3 x ULN vi. Total Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL) vii. The patients need to have a forced expiratory volume (FEV1) ≥ 1.2 liters or >40% predicted value viii. INR/APTT within normal limits;
6. All patients are notified of the investigational nature of this study and signed a written informed consent in accordance with institutional and national guidelines, including the Declaration of Helsinki prior to any trial-related intervention;
7. Patients aged > 18 years;
8. Women of childbearing potential, including women who had their last menstrual period in the last 2 years, must have a negative serum or urine pregnancy test within 7 days before randomization.

   All sexually active men and women of childbearing potential must use an effective contraceptive method (two barrier methods or a barrier method plus a hormonal method) during the study treatment and for a period of at least 12 months following the last administration of trial drugs;
9. Patient capable of proper therapeutic compliance and accessible for correct follow-up;
10. Measurable or evaluable disease (according to RECIST 1.1 criteria).

Exclusion Criteria:

1. All patients carrying activating mutations in the TK domain of EGFR or any variety of alterations in the ALK gene.
2. Patients with active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement or unexpected conditions of recurrence in the absence of an external trigger are allowed to be included.
3. Patients with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of randomization. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
4. Patients with a history of interstitial lung disease cannot be included if they have symptomatic ILD (Grade 3-4) and/or poor lung function. In case of doubt please contact trial team.
5. Patients with other active malignancy requiring concurrent intervention and/or concurrent treatment with other investigational drugs or anti-cancer therapy
6. Patients with previous malignancies (except non-melanoma skin cancers, and the following in situ cancers: bladder, gastric, colon, endometrial, cervical/dysplasia, melanoma, or breast) are excluded unless a complete remission was achieved at least 2 years prior to study entry AND no additional therapy is required during the study period.
7. Any medical, mental or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or understand the patient information
8. Patients who have had prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways
9. Patients with positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection
10. Patients with known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
11. Patients with history of allergy to study drug components excipients
12. Women who are pregnant or in the period of breastfeeding
13. Sexually active men and women of childbearing potential who are not willing to use an effective contraceptive method during the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the major pathologic response (MPR) | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 45 months
  The major pathologic response is defined as less than 10% tumor cells in the pathologically resected specimen

SECONDARY OUTCOMES:
pathologic complete response | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 45 months
  defined as no tumor cells observed in pathologically resected specimens
Resectable rate | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 45 months
  defined as the number of patients who underwent surgical resection/the number of randomized patients in each group
Disease-free survival | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 45 months
  defined as the interval from the surgery to the observation of confirmed disease recurrence

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat sen University cancer center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhao ZR, Yang CP, Chen S, Yu H, Lin YB, Lin YB, Qi H, Jin JT, Lian SS, Wang YZ, You JQ, Zhai WY, Long H. Phase 2 trial of neoadjuvant toripalimab with chemotherapy for resectable stage III non-small-cell lung cancer. Oncoimmunology. 2021 Oct 25;10(1):1996000. doi: 10.1080/2162402X.2021.1996000. eCollection 2021. PMID 34712513